CLINICAL TRIAL: NCT05583630
Title: Ligament Tension Measurement in Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Xu Zhihong, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2022-LCYJ-MS-23
Record Dates: First submitted 2022-09-15; First posted 2022-10-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Knee Arthropathy
Keywords: ligament tension, knee arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ligament tension measurement group: All participants will receive ligament tension measurement by the tension device during operation
  Interventions: Device: A gap plate with the function of knee joint pressure detection

INTERVENTIONS:
Device: A gap plate with the function of knee joint pressure detection — A gap plate can measure knee joint pressure by tension sensor. This is a part of routine medical care.

SUMMARY:
1. To develop a new type of knee joint pressure detection device and demonstrate its feasibility
2. To analyze individual differences of knee ligament tension using the new device and explore the influencing factors of ligament tension
3. To explore the correlation between knee ligament tension and postoperative knee function

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving primary knee arthroplasty

Exclusion Criteria:

* Patients having had a surgery history of the ipsilateral knee

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population are those receiving primary knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Ligament tension | During operation
  Measure the medial and lateral ligament tension of the operative knee at different flexion angle
Pre-operative knee function | 1day before operation
  Assess the knee function using AKS (The American knee society, 0~200, higher scores mean a better outcome) scale before operation
Post-operative knee function | The 3rd day after operation
  Assess the knee function using AKS scale at the 3rd day post-operation
Post-operative knee function | The 6th week after operation
  Assess the knee function using AKS scale at the 6th week post-operation
Post-operative knee function | The 3rd month after operation
  Assess the knee function using AKS scale at the 3rd month post-operation
Post-operative knee function | The 12th month after operation
  Assess the knee function using AKS scale at the 12th month post-operation

SECONDARY OUTCOMES:
Pre-operative infection test | 1day before operation
  Include C-reactive protein (CRP)
Pre-operative infection test | 1day before operation
  Include Erythrocyte Sedimentation Rate (ESR)
Pre-operative infection test | 1day before operation
  Include white blood cell
Post-operative infection test | The 1st day after operation
  Include CRP
Post-operative infection test | The 1st day after operation
  Include ESR
Post-operative infection test | The 1st day after operation
  Include white blood cell

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Xu, Doctor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available by consulting the principal investigator